CLINICAL TRIAL: NCT02295644
Title: Immediate Effect of Ultrasound Therapy on Bilateral Masseter Myalgia: Randomized Single Blinded Investigational Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, W.D.McCall, Jr., Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUNYBuffalo
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Therapeutic ultrasound
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: 0.4 Watts/Sq cm 50% Duty cycle (Experimental): 0.4 Watts/Sq cm 50% Duty cycle Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1 (MegaHertz) MHz, 5 minutes
  Interventions: Device: Ultrasound Sonicator 740
- B: 0.4 Watts/Sq cm 100% Duty cycle (Experimental): 0.4 Watts/Sq cm 100% Duty cycle Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1 MHz, 5 minutes
  Interventions: Device: Ultrasound Sonicator 740
- C: 0.8 Watts/Sq cm 50% Duty cycle (Experimental): 0.8 Watts/Sq cm 50% Duty cycle Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1 MHz, 5 minutes
  Interventions: Device: Ultrasound Sonicator 740
- D: 0.8 Watts/Sq cm 100% Duty cycle (Experimental): 0.8 Watts/Sq cm 100% Duty cycle Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1 MHz, 5 minutes
  Interventions: Device: Ultrasound Sonicator 740

INTERVENTIONS:
Device: Ultrasound Sonicator 740 — Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes

SUMMARY:
Introduction. Temporomandibular disorders (TMD) are a group of conditions that are multifactorial in nature, and it primarily presents with symptoms of pain and decreased functional capacity. Therapeutic ultrasound is a method of physical therapy that has shown clinically to provide immediate relief of pain in patients with different musculoskeletal disorders. In this study, for the purpose of immediate management of painful masticatory muscle and tissues, the investigators attempt to understand the mechanism of therapeutic ultrasound by exploring the physiologic changes peripherally and centrally. In addition, the investigators aim to determine if there is a dose response relationship between two different intensities (0.4 W/cm2 and 0.8 W/cm2) and between two sets of duty cycles (50% and 100%). A third purpose is to determine if therapeutic ultrasound applied to the masseter muscle is capable of eliciting segmental effects in the temporalis muscle. Methods. A total of 28 adult females with bilateral myalgia according to Diagnostic criteria for TMD (DC/TMD) will be recruited for this investigational trial. Each subject will be randomly allocated to one of the four ultrasound intervention groups each of which has different settings. Using Sonicator®740, therapeutic ultrasound intervention will be performed on both masseters for five minutes on each side of the face. A template will be used to confine the borders of the muscle and to determine the sites for the repeated outcome measures. Outcome parameters of: self-reported pain scale, pressure pain threshold, electromyographic muscle amplitudes and intraoral muscle temperatures will be measured for masseter and temporalis muscles on each side of the face, and will be assessed at baseline and after intervention on each side.

DETAILED DESCRIPTION:
The "Brief Summary" above encompasses the detailed description.

ELIGIBILITY:
Inclusion Criteria:

* Adult females who have bilateral myalgia based on Diagnostic Criteria for TMD (DC-TMD) criteria and current pain intensity (≥4 out of 10, where 0 is no pain and 10 is the worst pain ever) on both sides.

Exclusion Criteria:

* Those who have a history or were diagnosed with systemic musculoskeletal disorders or rheumatologic diseases (e.g. fibromyalgia, muscular atrophy).
* Certain conditions such as neoplasms or fractures.
* Neuropathies or neurological disorders.
* Participants who are currently taking muscle relaxants or analgesics.
* Those who have undergone any form of physical therapy within the last 60 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willard McCall, Principal Investigator — State University of New York at Buffalo
Locations (1):
- School of Dental Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- A (0.4W/Square Centimeter, 50%): 0.4 Watts/Sq cm 50% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
- B (0.4W/Square Centimeter, 100%): 0.4 Watts/Sq cm 100% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
- C (0.8W/Square Centimeter, 50%): 0.8 Watts/Sq cm 50% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
- D (0.8W/Square Centimeter, 100%): 0.8 Watts/Sq cm 100% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
Period: Overall Study
Arm/Group | A (0.4W/Square Centimeter, 50%) | B (0.4W/Square Centimeter, 100%) | C (0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%)
Started | 7 (All groups were randomly allocated to subjects upon the start of their individual trials) | 7 (All groups were randomly allocated to subjects upon the start of their individual trials) | 7 (All groups were randomly allocated to subjects upon the start of their individual trials) | 7 (All groups were randomly allocated to subjects upon the start of their individual trials)
Completed | 7 | 7 | 6 | 5
Not Completed | 0 | 0 | 1 | 2
Not completed — Did not meet inclusion criterion | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: One in group C and two in group D did not meet inclusion criterion of reporting current pain intensity of ≥4 on the Diagnostic Criteria for TMD.
Groups:
- A(0.4W/Square Centimeter, 50%): 0.4 Watts/Sq cm 50% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
- B(0.4W/Square Centimeter, 100%): 0.4 Watts/Sq cm 100% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
- Total: Total of all reporting groups
Arm/Group | A(0.4W/Square Centimeter, 50%) | B(0.4W/Square Centimeter, 100%) | C (0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%) | Total
Number analyzed (Participants) | 7 | 7 | 6 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 6 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 5 | 25
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Self Report of Pain
Description: Pain intensity measurement scale from 0 to 10, 0 is no pain, 10 is the worst pain ever
Time Frame: Immediately before and after the intervention, difference used.
Measure: Mean (Standard Deviation); unit: Scores on pain intensity scale
Arm/Group | A (0.4W/Square Centimeter, 50%) | B (0.4W/Square Centimeter, 100%) | C (0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%)
Number analyzed (Participants) | 7 | 7 | 6 | 5
Scores on pain intensity scale | -.86 (1.4) | -2.0 (.87) | -1.4 (1.1) | -1.3 (1.4)
Statistical Analysis 1: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = 0.17, ANOVA — Interaction test of duty cycle and intensity for self reported pain score
Statistical Analysis 2: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = 0.14, ANOVA — Main effect of duty cycle on self reported pain score
Statistical Analysis 3: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = 1.0, ANOVA — Main effect of intensity on self reported pain score

2. Primary Outcome: Pressure Pain Threshold of the Masseter Muscle
Description: Measuring pressure pain threshold using digital algometer
Time Frame: Immediately before and after the intervention, difference used.
Measure: Mean (Standard Deviation); unit: Kpa/Cm^2
Arm/Group | A (0.4W/Square Centimeter, 50%) | B (0.4W/Square Centimeter, 100%) | C (0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%)
Number analyzed (Participants) | 7 | 7 | 6 | 5
Kpa/Cm^2 | -2.64 (31.79) | 15.21 (5.75) | -5.12 (9.44) | -10.2 (12.04)
Statistical Analysis 1: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = .24, ANOVA — Main effect for duty cycle
Statistical Analysis 2: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = 0.019, ANOVA — Main effect for intensity
Statistical Analysis 3: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Interaction of intensity and duty cycle; Test type: Superiority or Other; p = 0.17, ANOVA

3. Primary Outcome: Intraoral Muscle Temperature
Description: Using digital thermometer on buccal mucosa, degrees celsius.
Time Frame: Immediately before and after the intervention, difference used.
Measure: Mean (Standard Deviation); unit: degrees Celsius, post minus pre
Arm/Group | A (0.4W/Square Centimeter, 50%) | B (0.4W/Square Centimeter, 100%) | C (0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%)
Number analyzed (Participants) | 7 | 7 | 6 | 5
degrees Celsius, post minus pre | .036 (.09) | .15 (.206) | .033 (.154) | .42 (.40)
Statistical Analysis 1: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Test type: Superiority or Other; p = 0.034, ANOVA — Main effect for duty cycle
Statistical Analysis 2: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Main effect for intensity; Test type: Superiority or Other; p = 0.475, ANOVA
Statistical Analysis 3: Comparison: A (0.4W/Square Centimeter, 50%) vs B (0.4W/Square Centimeter, 100%) vs C (0.8W/Square Centimeter, 50%) vs D (0.8W/Square Centimeter, 100%); Interaction of intensity and duty cycle; Test type: Superiority or Other; p = .178, ANOVA

ADVERSE EVENTS:
Time Frame: Throughout the trial of one hour.
Groups:
- C(0.8W/Square Centimeter, 50%): 0.8 Watts/Sq cm 50% Duty cycle
  Ultrasound Sonicator 740: Therapeutic ultrasound (Ultrasound Sonicator 740) used on masseter muscle, 1MHz, 5 minutes
Arm/Group | A(0.4W/Square Centimeter, 50%) | B(0.4W/Square Centimeter, 100%) | C(0.8W/Square Centimeter, 50%) | D (0.8W/Square Centimeter, 100%)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
Three subjects who met the inclusion criteria on recruitment (bilateral masseter pain of four or more) did not meet the criteria at the time of the experiment so were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No